CLINICAL TRIAL: NCT05058885
Title: Plasmodium Vivax Burden, Range and Transmission Among Duffy Negative Inhabitants in Cameroon.
Brief Title: Plasmodium Vivax Among Duffy Negative Population in Cameroon.
Acronym: VIBRANT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Dschang (Other)
Collaborators: Barcelona Institute for Global Health (Other); University of Yaounde 1 (Other)
Responsible Party: Principal Investigator, Dr Innocent Ali, Senior Lecturer, University of Dschang
Other Study IDs: TMA2020CDF-3171.
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Malaria, Vivax; Malaria,Falciparum; Malaria
Keywords: Serology,; Vivax; Malaria; Duffy-negative; Cameroon
MeSH Terms: conditions — Malaria, Vivax; Malaria, Falciparum; Malaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Finger-stick blood spots on Whatman n3 filter papers.

SUMMARY:
Although Plasmodium vivax (P. vivax), one of the five malaria species causing parasites, has the widest geographical distribution, it is rare in sub-Saharan Africa due to the absence of a red blood cell receptor (Duffy antigen) in black Africans. Duffy-negative individuals are, for the most part, therefore refractory to P. vivax infection and the Duffy-negative phenotype is found at highest frequencies in Africa, whereas it is relatively rare elsewhere. P. vivax has however, been observed as single infections in up to 5% of Duffy-negative febrile patients in one health facility in Dschang, a region of low malaria transmission in Western highlands of Cameroon. Whereas in the littoral South West and Southern forest of Cameroon characterised by high malaria transmission, areas, there are contrasting molecular evidence of human P. vivax infection. While important, the significance is limited from an epidemiological point of view, concerning the source, transmission, distribution range of P. vivax. There is thus a challenge in the true estimation of malaria burden, as well as the attributable parasite species in infections occurring in the low transmission areas of Western Cameroon. As a consequence, our understanding of the local epidemiology of malaria in Western Cameroon warrants formal investigation. The current proposal is a multi-centre observational study. Its purpose is to characterise the malaria species composition and particularly exposure and burden of P. vivax across malaria endemic settings in Cameroon. It will use multiplex serological methods based on quantitative suspension array on finger-stick blood samples collected from febrile patients of ages 1-100 during two malaria transmission seasons in different eco-climatic regions in Cameroon.

DETAILED DESCRIPTION:
Type of study:

The current proposal is a multi-centre observational study in different eco-climatic regions in Cameroon.

Study locations:

Dschang health district(Low transmission, highland) , Maroua (Sahel, high transmission) and Bertoua-Batouri (East region, forest, perennial transmission).

Study period:

The study will be conducted over a period of 36 months beginning from June, 2021.

Study population:

In each selected health facility, children 1 year and above, and adult of both gender will be eligible for participation.

Selection criteria: inclusion criteria, exclusion criteria.

Inclusion criteria:

1. Patient must be febrile (temperature >37.50 C or history of fever within 24 hours of arrival to the hospital)
2. Patient must be aged 1 year or older
3. Both males and females alike
4. The patient must be able to sign a consent/assent form
5. The patient must be seeking care and be suspected of malaria infection

Non-inclusion criteria:

1. Patient less than 1 year
2. Patient not having fever
3. Patient not being suspected of malaria infection

Exclusion criteria:

1. Eligible patient who refuses consent to study procedures
2. Patient withdraws consent before or during the start of study procedures
3. Patient, who, for any reason, refuses that sensitive data should not be processed.

6) Recruitment strategies for the study population

Sample size and justification:

This study is a cross sectional study that will determine a point estimate of the seroprevalence of parasite species, and in particular Plasmodium vivax in Cameroon. For this reason, we calculated the sample size based on an estimate of Plasmodium vivax in febrile patients as reported in a study in 2017((1)https://malariajournal.biomedcentral.com/articles/10.1186/s12936-017-1722-2), to get the highest power to calculate the sample population size for use in our study. Using the formula n = [DEFF*Np(1-p)]/ [(d2/Z21-α/2*(N-1)+p*(1-p)] in which DEFF=design effect=1, p =Hypothesised percentage frequency of outcome factor in the population=25%, from above study, d=confidence limit=5%, n=sample size, investigators calculated the for the study in three sites to be 867 or 300 per site, taking into consideration a refusal rate 4%. The software OpenEpi was used or the calculations (http://www.openepi.com/SampleSize/SSPropor.htm).The primary outcome is the spatial seroprevalence of Plasmodium vivax among febrile patients in the three epidemiological facies in Cameroon. For entomological component, WHO methods for Human landing catch (HLC) will be used to catch mosquitoes in 12-15 houses in each of four neighbourhoods over the periods corresponding to the beginning of malaria transmission, the peak malaria transmission and at the end of the malaria transmission season.

8) Sample collection procedure:

In each selected health facility, febrile individuals 1 year and above will be eligible for biological sample collection. Volunteers who have provided written informed consent/assent will have a finger prick sampling (approximately 500μl). Four Dried Blood Spots (DBS, Whatman 903 Protein Saver) will be prepared for immunological and molecular assays.

Serological analysis

Six Plasmodium antigens will be used to screen patient samples: two P.f antigens (Merozoite Surface Protein-1 19kD (MSP-1) and Apical Merozoite Antigen-1 (AMA-1), three P. vivax antigens (PvMSP-1 and PvAMA-1, pvRBPII), one P. malariae (PmMSP-1) and one P. ovale (PoMSP-1) selected on the basis of previous studies (20). Recombinant antigen will serve as a generic protein to assess immunoglobulin G (IgG) non-specific binding. Antigens for other species of malaria causing parasites are used in order to eliminate cross reacting sera and identify co-infections from pure P. vivax infections.

Data analysis and management.

Data Management:

Field data will be entered into a password-protected database designed for the study through hand held tablets at each study site. Primary data collection tool such as paper questionnaires will be stored in metal cupboards with access control maintained by the principal investigator of the study. Geographical location will be collected, but in the dataset, it will be perturbed as well, by replacing with other coordinates which will not distort the utility of the geolocation data and at minimum that the exact location of study participants is not discernable.

Data analysis

Data will be cleaned centrally by visual inspection for outliers. The primary study outcome for this will be the seroprevalence of P. vivax in the enrolled population of febrile patients in different geo-ecological regions of Cameroon. The Bayesian analytical framework using several different tools such as geographical positioning system, will be used to characterise the spatial seroprevalence across different ecologies using individual and geographical covariates in the model. The spatial software SaTScan will be used to identify clusters of antibody responses against each antigen. The spatial analysis will be run separately for each survey and spatial autocorrelation of clusters for each of the two survey time points assessed using Moran's I in ArcGIS software, as done previously (22). Age-adjusted antibody residuals from the regression model will be used for this analysis. Risk factors for P. vivax infection will be assessed using mixed effect logistic regression analysis with sampling site (health facility) considered a random effect variable. The Microsoft Excel suite as well as the latest version of STATA or R-package will be used as the statistical software.

Ethical considerations: potential risks, benefits, measures taken for data confidentiality and respect for the privacy of participants

This is a minimal risk study that has an ethical clearance renewal from the IRB of the Cameroon Baptist Convention health Services. This clearance will be renewed yearly until close of study from the National Ethics Committee for Human Health Research (CNERSH). No remuneration to participants will be made. Only de-identified datasets will be used for analysis. At the end of the study, all hard copy materials and the study key will be destroyed. This will follow local regulations that state a maximum of 15 years for data and 10 years for biological materials. The ethical committee requires that they be reached in case a study participant feels his/her rights are being violated. In all information sheets (of which the participant will have a copy), the mobile phone number of the responsible contact of the ethical committee will be mentioned.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be febrile (temperature >37.50 C or history of fever within 24 hours of arrival to the hospital)
* Patient must be aged 1 year or older
* Both males and females alike
* The patient must be able to sign a consent/assent form
* The patient must be seeking care and be suspected of malaria infection

Exclusion Criteria:

* Eligible patient who refuses consent to study procedures
* Patient withdraws consent before or during the start of study procedures
* Patient, who, for any reason, refuses that sensitive data should not be processed.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: n each selected health facility, children 1 year and above, and adult of both gender will be eligible for participation. Those who provide written consent/assent will be recruited in the study and be seen only once. All eligible and consenting individuals including women, children and other vulnerable persons will be part of the study as risk of infection with Plasmodium vivax, and malaria in general is the same for everyone living in Cameroon. Appropriate (ethical) measures will be taken when including vulnerable persons and children
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of P. vivax exposed patients in different eco-climatic settings in Cameroon | June 2022-June 2023
  A cut-off for seropositivity will be determined based on the mean of log MFI values plus three standard deviations of the seronegative controls. Separate cut-off values will be generated for each of the studied antigens. By so doing, participants will be classified as seropositive or seronegative depending on whether their antibody levels lie above or below the cut-off values. The seroprevalence will be calculated for each antigen, as the proportion of seropositive individuals of the total study population, per study site, and overall.
Species ratio among febrile patients infected with Plasmodium spp in geo-ecological regions of Cameroon. | June 2022-June 2023
  This will be defined as the ratio of each of identified species by serology to the total species observed for the particular region and, if required, for the overall study sites.

SECONDARY OUTCOMES:
Vector type, abundance, infectivity and anthropophily | June 2022-December, 2023.
  This outcome will include a determination of the vector type and infectivity of the mosquitoes with Plasmodium as determined by published molecular methods.
Entomological innoculation rate of vivax mosquitoes | June 2022-December, 2023.
  Established methods will be used to determine the number of infective bites per person and per year.

CONTACTS AND LOCATIONS:
Locations (1):
- Dschang Health District, Dschang, West Region, Cameroon